CLINICAL TRIAL: NCT01870986
Title: Phase 1, Double Blind, Randomized, Parallel-Group, Single-Dose, 3-Arm, Comparative Pharmacokinetic Study Of PF-06410293 and Adalimumab Sourced From US And EU Administered To Healthy Subjects
Brief Title: Study Of PF-06410293 And Adalimumab In Healthy Subjects (REFLECTIONS B538-01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B5381001; REFLECTIONS B538-01
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Phase 1; PK; adalimumab; Single-dose; Immunology; Bioequivalence; Biosimilarity; Similarity.
MeSH Terms: interventions — PF-06410293; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): PF-06410293
  Interventions: Biological: PF-06410293
- B (Active Comparator): Adalimumab-EU
  Interventions: Biological: Humira (adalimumab-EU)
- C (Active Comparator): Adalimumab-US
  Interventions: Biological: Humira (adalimumab-US)

INTERVENTIONS:
Biological: PF-06410293 — 40 mg/0.8 mL administered by sub-cutaneous injection with a single-use prefilled syringe.
  Other Names: adalimumab-Pfizer
  Arms: A
Biological: Humira (adalimumab-EU) — 40 mg/0.8 mL administered by sub-cutaneous injection with a single-use prefilled syringe.
  Other Names: adalimumab (European Union)
  Arms: B
Biological: Humira (adalimumab-US) — 40 mg/0.8 mL administered by sub-cutaneous injection with a single-use prefilled syringe.
  Other Names: adalimumab (United States)
  Arms: C

SUMMARY:
This healthy volunteers study will evaluate 210 subjects who will receive a single sub-cutaneous dose of PF-06410293 or adalimumab (United States) or adalimumab (European Union). This study will involve sampling and pharmacokinetics evaluation of drug levels following administration of PF-06410293 and the licensed adalimumab products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (non-childbearing potential). Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure, pulse, ECG, and laboratory testing.

Exclusion Criteria:

* Evidence or history of clinically significant infectious, hematological, renal, endocrine, pulmonary gastrointestinal, cardiovascular, hepatic psychiatric, neurologic, autoimmune, or allergic disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Day 1 - Day 43
Area Under the Curve From Time Zero to Last Time Point with Quantifiable Concentration (AUClast) | Day 1 - Day 43
Area under the Concentration-Time Curve (AUC) from Time Zero extrapolated to infinity (AUCInf) | Day 1 - Day 43

SECONDARY OUTCOMES:
Incidence of anti-adalimumab antibodies (ADA) and neutralizing antibodies (Nab) | Day 1 - Day 71
Time to Reach Maximum Observed Serum Concentration (Tmax) | Day 1- Day 43
Area under the Concentration-Time Curve (AUC) time Zero to 2 weeks after Dosing | Day 1- Day 43
Systemic Clearance (CL) | Day 1- Day 43
Serum Decay Half-Life (t1/2) | Day 1- Day 43
  Serum decay half-life is teh time for the serum concentration to decrease by one half

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, New Haven, Connecticut, United States
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5381001&StudyName=Study%20Of%20PF-06410293%20And%20adalimumab%20In%20Healthy%20Subjects%20%28REFLECTIONS%20B538-01%29